CLINICAL TRIAL: NCT05044533
Title: Evaluating QUAlity of Life of AF Patients Following a Bleed (EQUAL-AF)
Brief Title: A Study Evaluating Quality of Life for Participants With Atrial Fibrillation (AF) Following a Bleed (EQUAL-AF)
Acronym: EQUAL-AF
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-770
Record Dates: First submitted 2021-09-10; First posted 2021-09-14 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
Keywords: BMS-562247; Atrial Fibrillation; Oral Anticoagulant; Prospective Study; Quality of Life (QoL); United Kingdom
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with atrial fibrillation (AF) experiencing a bleed

SUMMARY:
The purpose of this observational study is to identify participants with both minor and major bleeds as a result of anticoagulant treatment for AF and evaluating their QoL through both primary and secondary care settings.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Adult patients (>= 18 years old)
* Patients who can understand all study information and literature to provide fully informed consent
* Atrial fibrillation (AF) as the primary diagnosis
* Having a major or minor bleed up to a maximum of 30 days prior to point of enrolment
* Receiving oral anticoagulation therapy for AF

Exclusion Criteria:

* Pregnant women
* Patients with active cancer
* Patients unable to consent for themselves
* Patient on concomitant antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18) who have Atrial fibrillation (AF) and are actively prescribed oral anticoagulant therapies (OATs) and have recently experienced bleeds, up to a maximum of 30 days prior to enrolment. No upper age limit will be applied, but patients must match all other inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Distribution of characteristics of AF participants: Quality of life (QoL) data | Up to 90 days
Distribution of characteristics of AF participants: Impact of the anticoagulation treatment | Up to 90 days

SECONDARY OUTCOMES:
Distribution of outcomes of AF participants: Timing of bleeding occurrence | Up to 90 days
Distribution of outcomes of AF participants: Nature of the bleed | Up to 90 days
Distribution of outcomes of AF participants: Current Bleeding treatment | Up to 90 days
Distribution of outcomes of AF participants: Location of bleed | Up to 90 days
Distribution of outcomes of AF participants: Documented cause of bleed | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Swansea, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm